CLINICAL TRIAL: NCT05806476
Title: Acute Caffeine Intake, Cognition and DNA Study
Brief Title: Caffeine, DNA and Cognition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Mary's University, Twickenham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: SMU_ETHICS_2021-22-319
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Function 1, Social
Keywords: cognition; caffeine; attention; memory; executive function; emotion recognition; genetics
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: the researchers prepared the caffeine and placebo capsules and someone outside the research team blinded them so that both the investigators and the participants were blinded. Identical opaque capsules were used for both caffeine and placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- C - C (Experimental): caffeine intake during the run-in days and caffeine intake on the experimental day
  Interventions: Dietary Supplement: caffeine
- C - P (Experimental): caffeine intake during the run-in days and placebo intake on the experimental day
  Interventions: Dietary Supplement: caffeine; Dietary Supplement: placebo
- P - P (Experimental): placebo intake during the run-in days and placebo intake on the experimental day
  Interventions: Dietary Supplement: placebo
- P - C (Experimental): placebo intake during the run-in days and caffeine intake on the experimental day
  Interventions: Dietary Supplement: caffeine; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: caffeine — 1.75mg / kg body mass of caffeine x 3 times a day during the run-in days and 3mg / body mass of caffeine once on the experimental days
  Arms: C - C; C - P; P - C
Dietary Supplement: placebo — 1.75mg / kg body mass of microcrystalline cellulose x 3 times a day during the run-in days and 3mg / body mass of microcrystalline cellulose once on the experimental days
  Arms: C - P; P - C; P - P

SUMMARY:
A study investigating the effects of acute caffeine intake on cognition based on genes associated with caffeine metabolism and physiological effect.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled crossover design that incorporates alternating periods of 'long-term' caffeine exposure and abstinence will be employed to investigate the inter-individual effects of caffeine on cognitive performance. The procedure that participants need to follow on each of the four weeks of the study is described in detail below.

1. Baseline visit: baseline questionnaire, anthropometry, familiarisation with study procedures and tasks. Participants will be supplied with week 1 supplementation (n= 18 capsules) and saliva vials (n= 6) for saliva sample collection. Participants will also be provided with decaffeinated coffee, tea and cocoa, depending on their preferences.
2. Days 1-6: placebo or caffeine capsules x 3 per day at 09.00, 11.00, and 15.00. Compliance with the caffeine and placebo supplementation will be assessed by a saliva sample at 17.00 every day for each of the days on long-term supplementation. Caffeine concentrations in blood and saliva correlate highly, and levels typically increase progressively during the day (due to intermittent consumption of caffeine beverages). The best single-sample bioassay of daily caffeine intake is provided by samples obtained in the late afternoon (James, 1994; James & Rogers, 2005).
3. Days 5 and 6: In preparation for the 'challenge' days and to control for environmental factors which have been shown to affect inducibility of CYP1A2 enzyme, participants will be asked to abstain from alcohol for 48 h and avoid strenuous exercise for 24 h before the trials and avoid consumption of cruciferous foods (broccoli and Brussels sprouts) (Gunes & Dahl, 2008). Finally, participants will be provided with diet diaries to record all food and beverages consumed during the 24 h before all four experimental trials.
4. Day 7 (Experimental day): Participants will be asked to present to the laboratory after an overnight fast and they will follow the procedure shown below:

09:00: Pre-supplementation saliva sample & cognitive tasks

09:30: Supplementation with 3 mg / kg body mass caffeine or placebo

10:30: First post-supplementation saliva sample & cognitive tasks

12:30: Second post-supplementation saliva sample & cognitive tasks

13:00: A meal containing of fruit juice or soft drink and a cheese sandwich

15:30: Third post-supplementation saliva sample & cognitive tasks

Saliva samples will be taken upon arrival and 1, 3 and 6 h post-supplementation. The first sample will be taken to verify adherence to the requirement not to take their morning supplementation, thus be in caffeine abstinence, regardless of the study arm. It has been shown that 1 mg/kg of caffeine results in caffeine plasma levels of about 1 μg/ml and salivary caffeine concentration may be expected to be about 70% of plasma levels (Walther et al., 1983). Mean saliva caffeine levels below 1 μg / ml have been previously reported for overnight caffeine abstinence (Evans & Griffiths, 1999). Following caffeinated treatment, salivary caffeine levels will aid in determination of caffeine metabolism (Dodd et al., 2015).

The supplementation will be swallowed with water proportional to participant weight (3-ml/kg body mass). During the experimental days, participants will be asked to consume water ad libitum in their first trial and an equal volume in the subsequent trials. They will also be asked to avoid exercise between the trials.

The cognitive tasks will be performed on four time points: pre- and 1, 3 and 6 h post-supplementation. When using anhydrous caffeine in capsules, peak caffeine concentration usually occurs around 1 h post ingestion (Graham, 2001). Therefore, measuring caffeine metabolites for 1 h post-caffeine ingestion would mostly measure caffeine absorption and not metabolism, which is determined by CYP1A2 enzyme. Thus, studies investigating the effects of CYP1A2 genotypes on caffeine effects should focus on using protocols which last >1 h, since these effects may be more evident in events lasting longer than 1 h, where the metabolism of caffeine may have a more pronounced effect. It should also be noted that the half-life of caffeine is on average 4-6 h (Nehlig, 2018) in most adults and it is not yet known to what degree caffeine metabolism is altered between fast and slow metabolisers. Therefore, it is unknown at what time point there would be a large enough difference in the circulating levels of caffeine between fast and slow metabolisers to have a significant impact on the ergogenicity of caffeine (Southward et al., 2018). For this reason, we selected 3 different time points post-supplementation to complete the cognitive tasks: 1 h post-supplementation was selected to permit comparison with several previous caffeine studies, because it is the most frequently used time point to test cognitive performance post-supplementation in the literature (Carswell et al., 2020). We also added the 3 h and 6 h post-supplementation time points since they are within the average range of caffeine half-life and to investigate the differences in performance between 'fast' and 'slow' metabolisers. We hypothesise that those who metabolise caffeine faster would not maintain high saliva levels of caffeine throughout the 6 h event compared to those with a slower metabolism of caffeine.

At the end of each experimental day, participants will be supplied with the capsules for the following week, as well as the vials for saliva caffeine sampling.

Once provided, samples will be kept frozen at -20 °C until analysis. Salivary caffeine levels will be measured using the Enzyme Multiplied Immunoassay Technique (EMIT) by spectrophotometric method. The EMIT assay is a homogenous enzyme immunoassay intended for use in determining caffeine as a metabolite and will be preferred given that it is less invasive than using serum caffeine and has been shown reliable and reproducible (Tripathi et al., 2015). Serum caffeine levels greater than 30 μg / ml require dilution when analysed by EMIT assay.

ELIGIBILITY:
Inclusion Criteria:

1) adult males and females 18-65 years; 2) who habitually consume caffeine; 3) free from any known disease; 4) free from medication, including contraceptive pills; 5) without uncorrected vision issues, e.g., having myopia but not wearing eyeglasses or daltonism (colour blindness); 6) non-smokers (to avoid contributory effects of nicotine or other tobacco substances to caffeine effects or tolerance) and 7) non-pregnant or breastfeeding.

Exclusion Criteria:

1) individuals with a chronic medical condition, 2) pregnant or lactating women, 3) regularly taking medication, including contraceptive pills, 4) with uncorrected vision, 5) smokers, 6) individuals who habitually consume alcohol more than the publicly recommended upper safe limits (21 and 14 units per week for men and women, respectively) and 7) not providing written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-04-04 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Attention and psychomotor speed | 8 min online task on 4 timepoints (n=4) on all experimental days (n=4)
  Attention and psychomotor speed is assessed using the Psychomotor Vigilance Task (PVT). The reaction times to optical stimulus (red dot) on the screen, measured in milliseconds will be used as a measure.
Memory | 6 min online task on 4 timepoints (n=4) on all experimental days (n=4)
  Memory is assessed using the N-back letter task. The reaction times for correct answers (was the letter on the screen displayed one/two/three letters ago? Yes or No), measured in milliseconds will be used as a measure.
Emotion recognition | 4 min online task on 4 timepoints (n=4) on all experimental days (n=4)
  Emotion recognition is assessed using the Karolinska Directed Emotional Faces. The reaction times for correct answers (what emotion does the person on the picture show? Anger, Fear, Disgust, Happiness, Sadness, Surprise), measured in milliseconds will be used as a measure.
Executive function | 5 min online task on 4 timepoints (n=4) on all experimental days (n=4)
  Executive function is assessed using the Stroop colour and word task. The reaction times for correct answers (name the word and name the colour of the word), measured in milliseconds will be used as a measure.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - St Mary's University Twickenham, London, Lobdon
  - St Mary's University, London

IPD SHARING:
Plan to Share IPD: No
participants have signed a consent form which clearly states who the members of the research team are and that their data will not be shared with anyone outside the research group, as part of their personal data protection